CLINICAL TRIAL: NCT01314703
Title: Test for Preoperative Skin Preparations
Brief Title: Topical Antimicrobial Effectiveness Testing
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 371.1.02.15.11
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Results first posted 2012-08-31 (Estimated); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Antimicrobial Effectiveness
MeSH Terms: interventions — 2-Propanol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ChloraPrep One-Step — 10.5 ml applicator preoperative skin preparation
Drug: 70% isopropyl alcohol — 10.5 ml applicator
  Other Names: Positive control

SUMMARY:
The primary objective of this study is to measure the antimicrobial effectiveness of ChloraPrep one-Step.

ELIGIBILITY:
Inclusion Criteria:

* in good general health
* have skin within 6 inches of the test sites that is free of tattoos, dermatoses, abrasions, cuts, lesions or other skin disorders.

Exclusion Criteria:

* topical or systemic antimicrobial exposure within 14 days prior to Screening Day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Bashir, MD, Principal Investigator — Microbiotest
Locations (1):
- Microbiotest, Sterling, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: March 05-April 04, 2011. Location: Microbiotest,clinical study center
Pre-assignment Details: 35 subjects entered pre-screening phase.2 subjects withdrew consent prior to the Screen Visit.33 subjects completed screen baseline.3 subjects did not meet screen baseline criteria.30 subjects qualified for treatment.3 subjects were discontinued prior to treatment because the required number of treatment sites were met. 27 subjects were treated.
Groups:
- ChloraPrep and 70% Isopropyl Alcohol: All subjects received treatment with both the ChloraPrep and 70% Isopropyl Alcohol
Period: Overall Study
Arm/Group | ChloraPrep and 70% Isopropyl Alcohol
Started | 35
Signed Informed Consent | 35
Completed Screen Visit | 33
Completed Treatment Visit | 27
Completed Study | 27
Excluded Prior to Screening Baseline | 2
Non Qualified Bacterial Screening Counts | 3
Discontinued When Enrollment Completed | 3
Completed | 27
Not Completed | 8
Not completed — screen failure and closed enrollment | 8

BASELINE CHARACTERISTICS:
Groups:
- Group 1: All subjects received treatment with both the test article and the positive control
Arm/Group | Group 1
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12.7) [19 to 62]
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Efficacy Will be Measured by the Change (+/-) in Bacterial Count on the Skin 10 Minutes After a Single Application of Test Material Relative to the Baseline Bacterial Count.
Description: the measure of antimicrobial efficacy was calculated by subtracting the 10 minute post test material application bacterial recovery from the baseline bacterial recovery.
Time Frame: 10 minutes after single application of test material
Population: 27 subjects were treated with ChloraPrep on the abdomen and groin treatment sites. 26 of the 27 abdomen sites met the qualifying bacterial baseline count and were included in the analysis. 25 of the groin sites met the qualifying bacterial baseline count and were included in the analysis.
Measure: Mean (95% Confidence Interval); unit: log 10 colony forming units
Groups:
- ChloraPrep One Step, 10.5 mL Applicator: All subjects received single application of treatment with ChloraPrep One Step 10.5 mL Applicator on two treatment sites (abdomen and groin).
- 70% Isopropyl Alcohol, 10.5 mL Applicator: All subjects received single application of treatment with 70% Isopropyl Alcohol 10.5 mL Applicator on two treatment sites (abdomen and groin).
Arm/Group | ChloraPrep One Step, 10.5 mL Applicator | 70% Isopropyl Alcohol, 10.5 mL Applicator
Number analyzed (Participants) | 27 | 27
log 10 colony forming units
  10 minute abdomen | 2.8469 [2.6699 to 3.0238] | 2.5328 [2.3559 to 2.7097]
  10 minute groin | 4.038 [3.7438 to 4.3322] | 3.5295 [3.2353 to 3.8237]
Statistical Analysis 1: Comparison: ChloraPrep One Step, 10.5 mL Applicator; Hypothesis: ChloraPrep will exceed 3 log 10 reduction for the groin at 10 minutes and 2 log 10 reduction for the abdomen at 10 minutes. The 70% Isopropyl Alcohol was used as a positive control. All calculations were performed after taking the base-10 logarithm of the original values. The model was a mixed model Analysis of Variance (ANOVA); Test type: Superiority or Other; ANOVA; Mean Difference (Net) = 2.85, 95% CI 2-sided [2.66 to 3.02], Standard Error of Mean 0.089 — ChloraPrep 10 minute abdomen
Statistical Analysis 2: Comparison: ChloraPrep One Step, 10.5 mL Applicator; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Mean Difference (Net) = 4.038, 95% CI 2-sided [3.74 to 4.33], Standard Error of Mean 0.149 — ChloraPrep 10 minute groin
Statistical Analysis 3: Comparison: 70% Isopropyl Alcohol, 10.5 mL Applicator; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Mean Difference (Net) = 2.53, 95% CI 2-sided [2.36 to 2.70], Standard Error of Mean 0.089 — 70%Isopropyl Alcohol 10 minute abdomen
Statistical Analysis 4: Comparison: 70% Isopropyl Alcohol, 10.5 mL Applicator; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Mean Difference (Net) = 3.53, 95% CI 2-sided [3.24 to 3.82], Standard Error of Mean 0.149 — 70% Isopropyl Alcohol 10 minute groin

ADVERSE EVENTS:
Time Frame: Study duration was approximately 21 days per study participant. Overall study duration was 28 days.
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No